CLINICAL TRIAL: NCT00004854
Title: The Safety and Efficacy of Adjunct Carvedilol in Children With Moderate Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Diagnostic
Other Study IDs: NCRR-M01RR00036-5073; M01RR000036 (NIH)
Record Dates: First submitted 2000-03-08; First posted 2000-03-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Heart Diseases
Keywords: moderate heart failure
MeSH Terms: conditions — Heart Diseases | interventions — Carvedilol

INTERVENTIONS:
Drug: Carvedilol

SUMMARY:
We would like to see if using Carvedilol in adjunct with Ace inhibitors will increase ejection fraction of the heart under echo. All interpretation of data will be sent to Boston Children's Hospital to be reviewed, which is the primary research center in this study. There are 5 hospitals participating in this study. The population targeted are children with moderate heart failure and must be on Ace inhibitors at the time of enrollment. Our outcome after placing them on Carvedilol is to change their ejection fraction on echo. The patients will be seen every 1-2 weeks, while we will titrate their medication to a maintenance dose. Secondary outcome is to increase quality of life, exercise tolerance and decrease their symptom scores as noted on their questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Etiology of heart failure in Group 1 or Group 2
* Moderate heart failure as evidenced by ventricular shortening fraction <= standard deviations below the mean, or ejection fraction <= 40% d) documented shortening fraction or ejection fraction that meet criteria for greater than 3 months
* Standard medical therapy include ACE inhibitors plus or minus diuretics plus or minus digoxin; all efforts will made to maximize therapy prior to entry. Medication doses must be stable for 3 months prior to entry
* Willingness to comply with followup testing

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States